CLINICAL TRIAL: NCT06904183
Title: Lenvatinib, Sintilimab, and Drug-Eluting Beads Transarterial Chemoembolization With or Without Hepatic Arterial Infusion Chemotherapy for Hepatocellular Carcinoma >7 cm With Portal Vein Tumor Thrombus: A Multicenter, Randomized Controlled Trial
Brief Title: Lenvatinib, Sintilimab, and DEB-TACE With/Without HAIC for HCC >7 cm With PVTT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Affiliated Hospital of Guangdong Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Huizhou Municipal Central Hospital (Other); Jieyang People's Hospital (Other); Guangzhou Development District Hospital (Unknown); First People's Hospital of Foshan (Other); Anqing Municipal Hospital (Other); Jinan University Affiliated Shunde Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIIR-25
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: hepatocellular carcinoma; lenvatinib; transarterial chemoembolization; drug-eluting bead; hepatic arterial infusion chemotherapy; portal vein tumor thrombosis; sintilimab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEN+SIN+DEB-TACE+HAIC (Experimental): Patients will receive the combination treatment of LEN+SIN+DEB-TACE+HAIC.
  Interventions: Combination Product: LEN+SIN+DEB-TACE+HAIC
- LEN+SIN+DEB-TACE (Active Comparator): Patients will receive the combination treatment of LEN+SIN+DEB-TACE.
  Interventions: Combination Product: LEN+SIN+DEB-TACE

INTERVENTIONS:
Combination Product: LEN+SIN+DEB-TACE+HAIC — For DEB-TACE, superselective catheterization is performed and DEBs loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session. After each chemoembolization, the microcatheter is reserved at the main hepatic tumor-feeding artery. The FOLFOX-based regimen is intra-arterially administered. During follow-up, the treatment of DEB-TACE and/or HAIC will be repeated for viable tumors based on the evaluation of the follow-up laboratory and imaging examination.
  Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd and sintilimab 200mg I.V. q3w will be started with 7 days after the first DEB-TACE+HAIC.
  Arms: LEN+SIN+DEB-TACE+HAIC
Combination Product: LEN+SIN+DEB-TACE — For DEB-TACE, superselective catheterization is performed and DEBs loaded with pirarubicin is use for chemoembolization. The embolization end point was blood stasis of the tumor-feeding arteries. In order to reduce the risk of complications, the embolization end point was not achieved in the initial TACE but in the second or third TACE session. During follow-up, the treatment of DEB-TACE will be repeated for viable tumors based on the evaluation of the follow-up laboratory and imaging examination.
  Lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd and sintilimab 200mg I.V. q3w will be started with 7 days after the first DEB-TACE.
  Arms: LEN+SIN+DEB-TACE

SUMMARY:
This study is conducted to evaluate the efficacy and safety of lenvatinib plus sintilimab, transarterial chemoembolization (TACE) with drug-eluting beads (DEB-TACE) and hepatic artery infusion chemotherapy (HAIC) with FOLFOX regemen (LEN+SIN+DEB-TACE+HAIC) versus lenvatinib plus sintilimab and DEB-TACE (LEN+SIN+DEB-TACE) for large hepatocellular carcinoma (> 7cm) with portal vein tumor thrombosis (PVTT).

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized study to evaluate the efficacy and safety of LEN+SIN+DEB-TACE+HAIC compared with LEN+SIN+DEB-TACE for unresectable large HCC (>7cm) with PVTT.

320 patients with large HCC (> 7cm) and PVTT will be enrolled in this study. The patients will receive either Len+DEB-TACE+HAIC or Len+DEB-TACE using an 1:1 randomization scheme. In the LEN+SIN+DEB-TACE+HAIC arm, the microcatheter will be reserved at the main hepatic tumor-feeding artery after DEB-TACE and chemotherapy drugs (oxaliplatin, fluorouracil and leucovorin; FOLFOX-based regimen) will be intra-arterially administered though the microcatheter. DEB-TACE+HAIC treatments can be repeated based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. In the LEN+SIN+DEB-TACE arm, patients will be treated with DEB-TACE alone. TACE treatment can be repeated based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team. In both arms, lenvatinib 12mg (body weight ≥60kg) or 8mg (body weight <60kg) P.O. qd and sintilimab 200mg I.V. q3w will be started within 7 days after the first DEB-TACE+HAIC/DEB-TACE.

The primary end point of this study is time to progression (TTP). The secondary endpoints are tumor response (objective response rate and disease control rate), overall survival (OS), and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of HCC
* the largest intrahepatic lesion >7 cm
* presence of PVTT on imaging
* tumor recurrence after curative treatment (hepatectomy or ablation) is eligible for enrollment
* Eastern Cooperative Oncology Group performance status ≤1
* Child-Pugh class A/B
* adequate hematologic and organ function, with leukocyte count>3.0×10^9/L, neutrophil count>1.5×10^9/L, platelet count≥75×10^9/L, hemoglobin 85 g/L, alanine transaminase and aspartate transaminase≤5×upper limit of the normal, creatinine clearance rate≤1.5×upper limit of the normal; prothrombin time prolongation ≤4 seconds
* life expectancy of at least 3 months

Exclusion Criteria:

* accompanied with vena cava tumor thrombus
* central nervous system involvement
* previous treatment with TACE, HAIC, TAE, radiotherapy, or systemic therapy
* organ (heart and kidneys) dysfunction, unable to tolerate TACE or HAIC treatment
* history of other malignancies
* uncontrollable infection
* history of HIV
* history of organ or cells transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | 4 years
  The time from date of randomization until the first occurrence of disease progression (according to mRECIST).

SECONDARY OUTCOMES:
Objective response rate (ORR) | 4 years
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to mRECIST.
Disease control rate (DCR) | 4 years
  The proportion of patients with the best response of CR, PR, or stable disease (SD) according to mRECIST.
Overall survival (OS) | 5 years
  The time from date of randomization to death due to any cause.
Adverse Events (AEs) | 4 years.
  Number of patients with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kangshun Zhu, Dr., Study Chair — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No